CLINICAL TRIAL: NCT01681537
Title: A Phase I Study of Lenalidomide Plus Chemotherapy With Mitoxantrone, Etoposide, and Cytarabine for the Reinduction of Patients With Acute Myelogenous Leukemia
Brief Title: Lenalidomide Plus Chemotherapy for AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Ballen, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-202
Record Dates: First submitted 2012-09-02; First posted 2012-09-10 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Lenalidomide; Mitoxantrone; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Lenalidomide and re-induction chemotherapy
  Interventions: Drug: Lenalidomide; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: Lenalidomide
Drug: Mitoxantrone
Drug: Etoposide
Drug: Cytarabine

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational combination of drugs. Phase I studies also try to define the appropriate dose of the investigational combination of drugs to use for further studies. "Investigational" means that the combination of drugs is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not approved this combination of drugs for AML. As part of this research study, you will take lenalidomide in combination with MEC. MEC are FDA approved chemotherapy drugs that are commonly used in the treatment of AML. Lenalidomide is approved by the FDA for patients with multiple myeloma, and some patients with myelodysplasia. Lenalidomide is considered investigational in this research study because it is not approved by the FDA for patients with AML.

Lenalidomide is a drug that affects the immune system, called an immunomodulatory drug or IMID. This drug is successful in the treatment of patients with multiple myeloma and some patients with myelodysplasia, a pre-leukemic condition. Other research studies suggest that lenalidomide may also be effective in patients with AML. Since we know that many patients who receive MEC chemotherapy alone do not have a prolonged remission (time free from leukemia), we are studying the addition of lenalidomide to MEC.

In this research study, we are looking for the highest dose of lenalidomide that can be given safely with MEC.

DETAILED DESCRIPTION:
After undergoing screening procedures to confirm that you are eligible to participate in the research study you will be admitted to the hospital. You will likely receive the majority of treatment on an inpatient basis. You will remain in the hospital for at least Days 4-8 and will be discharged at the discretion of your study doctor. It is likely that you will be hospitalized for several weeks due to the risk of infection after chemotherapy.

Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have relapsed or refractory AML, not everyone who participates in this research study will receive the same dose of the study drug. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses.

If you take part in this study you will be given a study drug-dosing calendar. There is only one cycle of treatment, which will be 28 days long. On Days 1 to 14 you will receive the lenalidomide orally. On Days 4-8 you will receive MEC chemotherapy: mitoxantrone by IV (intravenously, into your vein) over 30 minutes, etoposide by IV over one hour, and cytarabine by IV over one hour.

While on this study you will undergo a daily clinical exam for the first 14 days and then at least twice a week until your blood counts recover from treatment. A clinical exam consists of a physical exam, questions about your general health and specific questions about any problems that you might be having and any medications you may be taking. You will also undergo blood tests to assess your disease status and determine organ function level. This will happen daily for the first 14 days and then at least once a week (but up to 3 times per week) until your blood counts recover from treatment. Additionally a bone marrow aspirate/biopsy will be completed at the time of blood cell count recovery (usually between days 20 and 45) and as clinically indicated.

We would like to keep track of your medical condition for up to two years after your final dose of study drug. We would like to do this by getting in touch with you every 6 months to see how you are doing. Keeping in touch with you and checking your condition helps us look at the long-term effects fo the research study.

ELIGIBILITY:
Inclusion Criteria:

* Primary refractory disease following at least one cycle of induction therapy or first relapse or higher
* Must be registered into RevAssist program
* Able and willing to adhere to study schedule and other protocol requirements

Exclusion Criteria:

* Pregnant or breastfeeding
* Known hypersensitivity to thalidomide or lenalidomide
* Known seropositive for HIV
* Have had myocardial infarction within 6 months of enrollment or NYHA Class III or IV heart failure
* Other serious medical conditions or psychiatric conditions
* Major surgery within 28 days prior to treatment
* Received investigational agent or cytotoxic chemotherapy (except hydroxyurea) within 2 weeks of study
* Acute promyelocytic leukemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety of lenalidomide plus conventional chemotherapy for relapsed AML | 2 years
  Evaluation of the safety of lenalidomide in combination with conventional chemotherapy for relapsed acute myelogenous leukemia. Dose limiting toxicity is defined as a Grade IV rash or delayed neutrophil or platelet recovery beyond Day 45 after start of chemotherapy in the absence of disease

SECONDARY OUTCOMES:
Days to neutrophil recovery | 2 years
  Evaluation of neutrophil recovery (the first 3 days of ANC>500)
Complete Remission Rate | 2 years
  Evaluation of the complete remission rate and the complete remission rate without platelet recovery
Treatment-related mortality | 2 years
  Evaluation of the treatment-related mortality, the number of non-relapse related deaths in the first 45 days of starting treatment
Transfusion Support | 2 years
  Evaluation of transfusion support, the number of red blood cell and platelet transfusions needed in the first 45 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ballen, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts